CLINICAL TRIAL: NCT05214638
Title: Development and Application of Intelligent Assessment System of Longshi Scale
Status: Completed | Type: Observational
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20210812003-FS01
Record Dates: First submitted 2022-01-07; First posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Stroke; Disability Physical
Keywords: Stroke; Activities of Daily Living; Electronic Version
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assessed with the paper version of Longshi Scale first and then with electronic version
- Assessed with the electronic version of Longshi Scale first and then with the paper version

SUMMARY:
The purpose of this study was to verify convenience and feasibility of the novel intelligent Longshi assessment system to provide an accurate and convenient evaluation tool for stroke survivors.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Stroke survivors

      * age≥18 years
      * diagnosis of cerebral infraction or intracerebral hemorrhage
      * stable vital signs
      * willingness to participate in the study with informed consent
   2. Professional evaluators:

      * One to ten years of working experience
      * experience in rehabilitation scientific research or education related work for more than two years
      * association with Longshi Scale research
   3. Non-professional evaluators：

      * the family or caregiver of stroke survivors
      * ability to read and communicate
      * willingness to participate in the study with informed consent
2. Exclusion Criteria:

   1. Stroke survivors:

      * brain tumor, Parkinson's disease or active epilepsy within past three months
      * impaired cognitive functions
      * participation in any other clinical study
   2. Professional evaluators:

      * refusal to participate in the study
   3. Non-professional evaluators:

      * care for patients with serious mental health problems
      * refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors from the Department of Rehabilitation Medicine at Shenzhen Second People's Hospital are invited to participate in this study according to the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Consistency of the disability degree evaluated using the electronic version and the paper version of Longshi Scale | Within 48 hours
  Weighted kappa was used to determine the consistency of the disability degree evaluated using the electronic version and the paper version of Longshi Scale. Kappa value ranges from 0 to 1 and the thresholds for kappa reliability are as follows: poor (κ = 0.00-0.20), fair (κ= 0.21-0.40), moderate (κ = 0.41-0.60), good (κ = 0.61-0.80),and very good (κ = 0.81-1.00).

SECONDARY OUTCOMES:
Proportion of evaluators' preference | Within 48 hours
  After completing all the evaluations, each evaluator was asked to reveal their preferred version (paper version, electronic version or no preference). Chi-square test was used to compare the proportion of evaluators' preference.
Time required | Within 48 hours
  Time required in each section of electronic version and paper version of Longshi Scale.
Test-retest reliability of electronic version Longshi Scale | Within 48 hours after first evaluation
  Weighted kappa was used to determine test-retest reliability of electronic version Longshi Scale. Kappa value ranges from 0 to 1 and the thresholds for kappa reliability are as follows: poor (κ = 0.00-0.20), fair (κ= 0.21-0.40), moderate (κ = 0.41-0.60), good (κ = 0.61-0.80),and very good (κ = 0.81-1.00).

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

REFERENCES:
- [Derived] Xue K, Li W, Liu F, Liu X, Wong J, Zhou M, Cai C, Long J, Li J, Zhang Z, Hou W, Nie G, Wang Y. Evaluation of activities of daily living using an electronic version of the Longshi Scale in patients with stroke: reliability, consistency, and preference. BMC Med Inform Decis Mak. 2024 May 15;24(1):125. doi: 10.1186/s12911-024-02508-0. PMID 38750562